CLINICAL TRIAL: NCT01170507
Title: Magnitude of Changes in 25 OH Vitamin D3 Levels After Vitamin D3 Supplementation: A Randomized Controlled Study
Brief Title: Magnitude of Changes in 25 OH Vitamin D3 Levels After Vitamin D3 Supplementation
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No funding
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Muhammad Maher Hammami, Chairman, Department of Clinical Studies & Empirical Ethics, King Faisal Specialist Hospital & Research Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RAC 2101042
Record Dates: First submitted 2010-07-25; First posted 2010-07-27 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D3, 25 OH vitamin D3 level
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- vitamin D3 1000 IU (Active Comparator)
  Interventions: Drug: vitamin D3 1000 IU orally daily for 5 months
- Vitamin D3 3000 IU (Active Comparator)
  Interventions: Drug: vitamin D3 3000 IU orally daily for 5 months
- Vitamin D3 5000 IU (Active Comparator)
  Interventions: Drug: vitamin D3 5000 IU orally daily for 5 months
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo orally daily for 5 months

INTERVENTIONS:
Drug: vitamin D3 1000 IU orally daily for 5 months
  Arms: vitamin D3 1000 IU
Drug: vitamin D3 3000 IU orally daily for 5 months
  Arms: Vitamin D3 3000 IU
Drug: vitamin D3 5000 IU orally daily for 5 months
  Arms: Vitamin D3 5000 IU
Drug: Placebo orally daily for 5 months
  Arms: Placebo

SUMMARY:
Vitamin D deficiency is common world wide. 25 OH vitamin D level is the best indicator of vitamin D status. The determination of the appropriate dose of vitamin D supplement is essential for management of vitamin D deficiency as well as for designing vitamin D fortification programs. The increments in 25 OH vitamin D levels following various doses of vitamin D supplement for different genders, body weights, and starting 25 OH vitamin D level have not been well defined. The time course of depletion of repleted vitamin D stores is also not known.

The investigators plan to conduct a double blind randomized study on 9 cohorts to determine levels of 25 OH vitamin D following supplementation with different doses of vitamin D3 for 5 months and their withdrawal for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults living in Riyadh area who consume no more than one serving of milk/day, do not take vitamin supplement, habitually have less than 10 hr of sun exposure per week, don't suffer from granulomatous conditions, liver disease, or kidney disease, and don't take anticonvulsants, barbiturates, or steroids.
* Individuals with with total 25 OH vitamin D level exceeding 100 nmol/l will be excluded from the study. Individuals with 25 OH vitamin D levels less than 20 nmol/L will be excluded from the placebo arm.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Slope of 25 OH vitamin D3 level vs vitamin D3 dose | 5 months
  The primary endpoint is the slope of the dose (vitamin D3)- response (25 OH vitamin D3 level) curve for each cohort. The slope of the placebo group will be used to determine changes in 25 OH vitamin D3 levels that are not related to study intervention. The slope will be determined over 5 months.

SECONDARY OUTCOMES:
slope of vitamin D3 level vs vitamin D3 dose | 5 months
  slope of vitamin D3 level vs vitamin D3 dose over 5 months
incidence of hypercalcemia | 8 months
  incidence of hypercalcemia over 8 months
incidence of hypercalciuria | 8 months
  incidence of hypercalciuria over 8 months
slope of decline of 25 OH vitamin D3 level vs time | 3 months
  slope of decline of 25 OH vitamin D3 level vs time over 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad M Hammami, MD, PhD, Principal Investigator — King Faisal Specialist Hospital & Research Center
Locations (1):
- King Faisal Specialist Hospital & Research Center, Riyadh, Saudi Arabia